CLINICAL TRIAL: NCT04346277
Title: Compassionate Use Open-Label Anti-CD14 Treatment in Patients With SARS-CoV-2 (COVID-19)
Status: No longer available | Type: Expanded Access
Sponsor: Implicit Bioscience (Industry)
Responsible Party: Sponsor
Other Study IDs: COV02
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: COVID; ARDS, Human; Ards; SARS-CoV2
Keywords: coronavirus; acute lung injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Coronavirus Infections

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: IC14, a monoclonal antibody against CD14 — IC14 is a recombinant chimeric anti-human monoclonal antibody directed against human CD14. It recognizes both membrane-bound CD14 and soluble CD14.
  Other Names: anti-CD14

SUMMARY:
This protocol proposes to use IC14, a recombinant chimeric monoclonal antibody (mAb) recognizing human CD14, to block CD14-mediated cellular activation in patients early in the development of ARDS. The binding of IC14 to human CD14 prevents CD14 from participating in the recognition of PAMPs and DAMPs due to SARS-CoV-2 infection. The putative mechanism of action of IC14 in ARDS is blockade of PAMP and DAMP interactions with CD14, thus attenuating the inflammatory cascade that leads to increased endothelial and epithelial permeability and injury resulting in alveolar injury and fluid accumulation characteristic of ARDS.

IC14 is a chimeric monoclonal antibody that binds to CD14 with high affinity and inhibits signaling via membrane and soluble CD14. Blocking CD14 with IC14 treatment in normal volunteers strongly inhibits systemic inflammation in response to bacterial endotoxin (LPS). University of Washington conducted a small NIH-funded pilot trial of IC14 treatment in 13 patients with ARDS, which suggested that IC14 treatment reduced alveolar inflammation and decreased BAL cytokines. IC14 was also the subject of IND 105803 for a phase 2 study of ARDS from all causes which we propose to revise for the COVID-19 indication.

A dosing regimen for IC14 with favorable pharmacokinetics supporting once daily intravenous dosing has been defined, making this an acceptable treatment for hospitalized patients. Two pharmacodynamic biomarkers can be used that are related to CD14, measurements of sCD14 (serum at baseline; urine at baseline and follow up) as well as a CD14 fragment (sCD14-ST; presepsin). A CD14 target engagement assay is available.

Therefore, because of the central role of CD14 in the amplification of lung inflammatory responses leading to severe lung injury and the safety record of IC14 in humans, we propose to have an open-label protocol to test the safety and potential efficacy of IC14 treatment in preventing the progression of severe respiratory disease in patients hospitalized with COVID-19.

DETAILED DESCRIPTION:
This is a compassionate use open label program in patients hospitalized with pulmonary complications of SARS-CoV-2 infection who will receive IC14 at a dosage of 4 mg/kg on Day 1, then 2 mg/kg once daily on Days 2-4. Patient monitoring will be for a total of up to 28 days if the patient is still hospitalized.

Screening/baseline assessments and initiation of the first IC14 administration will occur within 48 hours after meeting inclusion criteria. IC14 should be administered at approximately 24-hr intervals beginning from the start time of the first IC14 administration (Day 1).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and able to give informed consent
2. Age 18-70 years
3. Presence of a SARS-CoV-2 infection documented by nasopharyngeal swab positive by RT-PCR testing or history of positive test
4. Radiologic findings compatible with diagnosis of SARS-CoV-2 pulmonary infection
5. Hypoxemia as defined by any of the following:

   1. SpO2 ≤92% on room air
   2. Requirement for >2L O2 per standard nasal cannula
   3. PaO2/FiO2<300 if on high-flow nasal cannula
6. Women of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

A patient fulfilling any of the following criteria is to be excluded from enrollment in the study:

1. Intubation
2. Do-not-attempt resuscitation (DNAR) / do not intubate status
3. Anticipated survival <48 hours
4. Anticipated survival <28 days due to pre-existing medical condition
5. Significant pre-existing organ dysfunction

   1. Lung: Currently receiving home oxygen therapy as documented in medical record
   2. Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record
   3. Renal: Chronic renal failure requiring renal replacement therapy
   4. Liver: Severe chronic liver disease defined as Child-Pugh Class C
6. Pre-existing, ongoing immunosuppression

   1. Solid organ transplant recipient
   2. Chronic high-dose corticosteroids (equivalent to >20 mg/prednisone/day for >14 days in the last 30 days)
   3. Oncolytic drug therapy within the past 14 days
   4. Known HIV positive with CD4 count <200 cells/mm3
7. Current treatment with Enbrel® (etanercept), Remicade® (infliximab), Humira® (adalimumab), Cimzia® (certolizumab), or Simponi® (golimumab), Kineret® (anakinra), Arcalyst® (rilonacept), or other potent immunosuppressant
8. Pregnancy
9. History of hypersensitivity or idiosyncratic reaction to IC14

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Scientific Institute, Vita-Salute San Raffaele University, Milan, Italy